CLINICAL TRIAL: NCT03953989
Title: A Pilot Study Assessing the Effects of Ranolazine on Coronary Microvascular Dysfunction in Patients With Hypertrophic Cardiomyopathy
Brief Title: Effects of Ranolazine on Coronary Microvascular Dysfunction in Patients With Hypertrophic Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Principal Investigator, Prof. Paolo G Camici MD FACC, Professor of Cardiology, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCMRanIT001
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: HCM - Hypertrophic Non-Obstructive Cardiomyopathy
MeSH Terms: interventions — Ranolazine

STUDY DESIGN:
Intervention Model Description: A pilot study, one center, open, non-controlled, one group pre-post treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hypertrophic cardiomyopathy (Experimental): Thestudy is articulated into Screening visit plus other 3 visits. One visit (V2 ) for dose titration. V0 screening eligibility, consent, Medical History, physical examination, BP, ECG, Echocardiography, Biochemistry (haematology, electrolytes, glycaemia, ALS and bilirubin, creatinine and urine-analysis) V1 Baseline PET scan, physical examination, vital signs, and drug supply (500 mg bid).
  V2 physical examination, safety check, biochemistry, drug compliance and up-titration (750 mg bid), drug supply.
  V3 (2 months)safety check ,drug supply, drug compliance V4 (4 months, end of treatment) repeat PET scan, physical examination, BP, ECG, drug compliance, safety.
  Drug of the study Ranolazine PR (prolonged-release) 500 mg 1 tablet bis in die and 750 mg 1 tablet bis in die
  Interventions: Drug: Ranolazine PR (prolonged-release) 500 mg 1 tablet bis in die and 750 mg 1 tablet bis in die

INTERVENTIONS:
Drug: Ranolazine PR (prolonged-release) 500 mg 1 tablet bis in die and 750 mg 1 tablet bis in die — Patients enrolled in the study, at the end of the titration phase will be treated with ranolazine 750 mg or 500 mg, 1 oral tablet twice a day for 4 months on top of standard of care treatment
  Other Names: Ranexa

SUMMARY:
To demonstrate the efficacy of ranolazine in improving coronary microvascular and diastolic dysfunction in patients affected by HCM evaluating changes in maximum (i.e. during dipyridamole-induced coronary vasodilatation) myocardial blood flow (MBF) measured by PET at baseline and after 4 months of treatment with ranolazine in patients with non obstructive HCM.

DETAILED DESCRIPTION:
This pilot study aimed at assessing the effects of treatment with ranolazine, on top of optimal standard medical therapy (according to international guidelines), on microvascular dysfunction using PET in patients with HCM.

Thirty months of enrolment are foreseen. Patients enrolled in the study, at the end of the titration phase will be treated with ranolazine 750 mg or 500 mg, 1 oral tablet twice a day for 4 months on top of standard of care treatment. Visit 0,1,2,3 may be performed 3 days before or 3 days after the planned date. Visit 4 and final PET scan may be performed 15 days before or 15 days after the planned date.

This is a superiority study. The sample size calculation is based on the ANOVA model, but the statistical analysis will be performed applying the ANCOVA model for the absence of data on the correlation between basal and end of study values of the primary variable studied. As previously reported (Camici et al. J Am Coll Cardiol 1991; 17:879-86) maximum (i.e. during dipyridamole stress) MBF is severely blunted in HCM (1.63±0.58 mL/min/g) compared to control subjects (2.99±1.06 mL/min/g). For the primary end-point of the study using a two-sided test at 5% significance level, with a power of 90% and a SD of ± 0.7 mL/min/gr, in order to detect a change of 0.5 mL/min/gr in maximum MBF before and after treatment, 24 patients valid per protocol are required.

ELIGIBILITY:
Inclusion Criteria:

* Male and female gender (females of childbearing potential must be using highly effective contraceptive precautions such as implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence or vasectomised partner);
* Females of childbearing potential or within two years from the menopause must have a negative urine pregnancy test;
* Patients which fulfill conventional echocardiographic criteria for the diagnosis of HCM: maximum LV wall thickness ≥ 15 mm;
* Patients aged > 18 years and < 80 years;
* Sinus rhythm accepted isolated Supraventricular and Ventricular Premature Beats (VPB);
* Absence of severe resting LV outflow tract obstruction (peak gradient ≤ 50 mmHg);
* Written informed consent prior to enrolment into the study;

Exclusion Criteria:

* Females of childbearing potential not using highly effective contraceptive precautions;
* Presence of known coronary artery disease (CAD);
* Presence of Chronic Obstructive Airways Disease;
* Asthma;
* Other causes of microvascular dysfunction including long-standing history of arterial hypertension, diabetes, uncontrolled dyslipidemia;
* Body mass index >32 kg/m2; < 17 kg/m2
* Overt LV systolic dysfunction with end-stage progression (LV-EF <50%);
* Concomitant administration of potent CYP3A4 inhibitors (e.g. itraconazole, ketoconazole, voriconazol, posaconazol, HIV protease inhibitors, clarithromycin, telithromycin, nefazodone);
* Patients treated with sotalol, dronedarone, class I antiarrhythmics (see appendix 4) or other QT-prolonging drugs; stable treatment with amiodarone is permitted;
* Patients with QTc (Bazett's formula) at baseline ≥ 450 ms males; ≥470 msec females;
* Any clinically relevant haematological or biochemical abnormality on routine screening, according to Investigator's judgment;
* Severe concurrent pathology, including terminal illness (cancer, AIDS, etc.);
* Severe renal impairment defined as GFR < 29 mL/min/1.73m2 or creatinine level > 2.5 mg/dL or BUN >60 mg/dL;
* Moderate or severe hepatic impairment or hepatic insufficiency defined as SGOT or SGPT > 2 times greater than normal upper limit of the local laboratory or total serum bilirubin > 1.5 times greater than normal upper limit of the local laboratory;
* Dementia, psychosis, alcoholism (>350 g ethanol/week) or chronic abuse of medicaments, drugs or psychoactive substances;
* Claustrophobia;
* Females who are pregnant or lactating;
* Conditions that in the Investigator's opinion may interfere with the study's execution or due to which the patient should not participate for safety reasons;
* Risk of poor patient cooperation;
* Participation in a clinical study ≤ 2 months before enrolment;
* Inability or unwillingness to issue the informed consent;
* Concomitant use of > 20 mg daily dose of Simvastatin during the study (in case of patients taking simvastatin > 20 mg daily, the switch to other statins not metabolized by the CYP3A4 could be considered);
* Concomitant use of Atorvastatin (> 80 mg daily)
* Concomitant use of > 1000 mg daily dose of metformin during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Myocardial Blood Flow during hyperemia ml/min/g | At baseline and after 4 months of treatment
  Change of near maximal hyperemic myocardial blood flow (MBF ml/min/g) after treatment with ranolazine of at least 0.5 ml/min/g. Myocardial perfusion measured with 13N-ammonia and positron emission tomography at rest and during hyperemia; Hyperaemic Myocardial Blood Flow (MBF) measured following i.v. dipyridamole (0.56 mg/Kg in 4 mins)
Coronary Flow Reserve (hyperaemic MBF /resting MBF = CFR). | At baseline and after 4 months of treatment
  Change of CFR after treatment with ranolazine for four months
Coronary resistance | At baseline and after 4 months of treatment
  Change of Resting coronary resistance (Mean Arterial Pressure rest/ MBF rest) and minimal (during hyperemia) coronary resistance (Mean arterial Pressure hyperemia/ MBF hyperemia)

SECONDARY OUTCOMES:
Symptoms | through 4 month of treatment
  Number of participants with absence of symptoms accountable for drug intolerability ,assessed through customized questionnaire. If symptoms are accountable for drug intolerability are referred, the patient will come back to 500 mg/bid.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Camici, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No